CLINICAL TRIAL: NCT02610556
Title: Concurrent Docetaxel Plus Cisplatin or Cisplatin Alone With Intensity-modulated Radiotherapy in High Risk Locregionally Advanced Nasopharyngeal Carcinoma: a Phase 2 Randomized Controlled Trial
Brief Title: Concurrent Docetaxel Plus Cisplatin or Cisplatin Alone With IMRT in High Risk Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-071-Dept. of RT
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: NPC; concurrent chemotherapy; docetaxel; cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — cisplatin-guanosine adduct; Docetaxel; SSRP1 protein, human; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TP plus IMRT (Experimental): Concurrent chemotherapy: TP - Docetaxel 60mg/m2, D1 and cisplatin 25 mg/m2, D1-3 every 3 weeks for 3 cycles; Radiation: Intensity-modulated radiotherapy
  Interventions: Drug: Docetaxel; Drug: Cisplatin 1; Radiation: Intensity-modulated radiotherapy
- DDP plus IMRT (Active Comparator): Concurrent chemotherapy: DDP - Cisplatin 100 mg/m2, D1 every 3 weeks for 3 cycles; Radiation: Intensity-modulated radiotherapy
  Interventions: Drug: Cisplatin 2; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Cisplatin 2 — Cisplatin 100 mg/m2, D1 every 3 weeks for 3 cycles
  Other Names: DDP
  Arms: DDP plus IMRT
Drug: Docetaxel — Docetaxel 60 mg/m2, D1 every 3 weeks for 3 cycles
  Other Names: T
  Arms: TP plus IMRT
Drug: Cisplatin 1 — Cisplatin 25 mg/m2, D1-3 every 3 weeks for 3 cycles
  Other Names: P
  Arms: TP plus IMRT
Radiation: Intensity-modulated radiotherapy — Intensity-modulated radiotherapy
  Other Names: IMRT

SUMMARY:
The investigators aim to evaluate the efficiency and toxicities of concurrent docetaxel and cisplatin with intensity-modulated radiotherapy in high risk locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Eligible patients are randomly assigned to receive intensity-modulated radiotherapy (IMRT) with concurrent chemotherapy of docetaxel plus cisplatin or cisplatin alone. IMRT is delivered with a total dose of 68 Gy or higher in 33 fractions to the primary tumor. Concurrent chemotherapy in the experimental arm consists of docetaxel 60 mg/m², D1 and cisplatin 25 mg/m², D1-3 every 3 weeks for 3 cycles. Concurrent chemotherapy in the control arm consists of cisplatin 100 mg/m², D1 every 3 weeks for 3 cycles.The primary endpoint is overall survival (OS), defined as time from randomization to the day of death from any cause. Secondary end points include failure-free survival (FFS), locoregional relapse-free survival (LRFS), distant metastasis-free survival (DMFS) and the incidence of grade 3 or higher acute toxicities. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologically confirmed non-keratinizing (WHO 1991) nasopharyngeal carcinoma.
* Tumor staged as T1N3M0, T2-3N2-3M0 or T4N0-3M0 (the 2010 UICC/AJCC staging system).
* Pretreatment EBV DNA ≥ 1500 copies/mL.
* Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4×10E9/L, hemoglobin ≥ 110g/L and platelet count ≥ 100×10E9/L.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and bilirubin ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min or creatinine ≤ 1.5×ULN.
* Patients must give written informed consent.

Exclusion Criteria:

* Prior malignancy, except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended radiotherapy volume).
* Prior radiotherapy, chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | two year

SECONDARY OUTCOMES:
failure-free survival | two year
distant metastasis-free survival | two year
locoregional relapse-free survival | two year
Number of participants with treatment-related acute adverse events as assessed by CTCAE v4.0 | up to two months

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Yun Xie, M.D., Principal Investigator — Sun Yat-sen University Cancer Center,Guangzhou, Guangdong, China
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang LN, Gao YH, Lan XW, Tang J, OuYang PY, Xie FY. Effect of taxanes-based induction chemotherapy in locoregionally advanced nasopharyngeal carcinoma: A large scale propensity-matched study. Oral Oncol. 2015 Oct;51(10):950-6. doi: 10.1016/j.oraloncology.2015.07.004. Epub 2015 Jul 21. PMID 26209065
- [Background] Xie FY, Zou GR, Hu WH, Qi SN, Peng M, Li JS. [Induction chemotherapy with docetaxel plus cisplatin (TP regimen) followed by concurrent chemoradiotherapy with TP regimen versus cisplatin in treating locally advanced nasopharyngeal carcinoma]. Ai Zheng. 2009 Mar;28(3):279-85. Chinese. PMID 19619443
- [Background] Tishler RB, Schiff PB, Geard CR, Hall EJ. Taxol: a novel radiation sensitizer. Int J Radiat Oncol Biol Phys. 1992;22(3):613-7. doi: 10.1016/0360-3016(92)90888-o. PMID 1346533
- [Background] Tishler RB, Geard CR, Hall EJ, Schiff PB. Taxol sensitizes human astrocytoma cells to radiation. Cancer Res. 1992 Jun 15;52(12):3495-7. PMID 1350755
- [Background] Komatsu M, Shiono O, Taguchi T, Sakuma Y, Nishimura G, Sano D, Sakuma N, Yabuki K, Arai Y, Takahashi M, Isitoya J, Oridate N. Concurrent chemoradiotherapy with docetaxel, cisplatin and 5-fluorouracil (TPF) in patients with locally advanced squamous cell carcinoma of the head and neck. Jpn J Clin Oncol. 2014 May;44(5):416-21. doi: 10.1093/jjco/hyu026. Epub 2014 Mar 30. PMID 24688084
- [Background] Inohara H, Takenaka Y, Yoshii T, Nakahara S, Yamamoto Y, Tomiyama Y, Seo Y, Isohashi F, Suzuki O, Yoshioka Y, Sumida I, Ogawa K. Phase 2 study of docetaxel, cisplatin, and concurrent radiation for technically resectable stage III-IV squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2015 Apr 1;91(5):934-41. doi: 10.1016/j.ijrobp.2014.12.032. PMID 25832686
- [Background] Higuchi K, Komori S, Tanabe S, Katada C, Azuma M, Ishiyama H, Sasaki T, Ishido K, Katada N, Hayakawa K, Koizumi W; Kitasato Digestive Disease and Oncology Group. Definitive chemoradiation therapy with docetaxel, cisplatin, and 5-fluorouracil (DCF-R) in advanced esophageal cancer: a phase 2 trial (KDOG 0501-P2). Int J Radiat Oncol Biol Phys. 2014 Jul 15;89(4):872-9. doi: 10.1016/j.ijrobp.2014.03.030. Epub 2014 May 24. PMID 24867539
- [Background] Chen X, Hong Y, Feng J, Ye J, Zheng P, Guan X, You X, Song H. Concurrent chemoradiotherapy comparison of taxanes and platinum versus 5-fluorouracil and platinum in nasopharyngeal carcinoma treatment. Chin Med J (Engl). 2014;127(1):142-9. PMID 24384440
- [Background] Baykara M, Buyukberber S, Ozturk B, Coskun U, Kaplan MA, Unsal DK, Dane F, Demirci U, Bora H, Benekli M; Anatolian Society of Medical Oncology. Efficacy and safety of concurrent chemoradiotherapy with cisplatin and docetaxel in patients with locally advanced nasopharyngeal cancers. Tumori. 2013 Jul-Aug;99(4):469-73. doi: 10.1177/030089161309900405. PMID 24326834
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714